CLINICAL TRIAL: NCT06366269
Title: Acupuncture as First-line Therapy for Patients With Interstitial Cystitis/Painful Bladder Syndrome
Brief Title: Acupuncture First for IC/BPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, David Sheyn, Physician, UHMG, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20240374
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Bladder Pain Syndrome; Interstitial Cystitis
Keywords: acupuncture; bladder pain syndrome; interstitial cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Acupuncture Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Group allocation will be masked to the care provider and investigators only while participants undergo the initial 6 weeks of treatment. Due to the nature of the intervention (acupuncture) participants are not able to be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Participants will receive instruction (verbal and written) on recommended changes to diet and urinary habits to treat bladder pain.
  They will complete six (6) weekly one hour acupuncture sessions followed by pelvic floor physical therapy.
  Interventions: Other: Acupuncture; Behavioral: Behavioral management; Other: Physical therapy
- Behavioral Management (Active Comparator): Participants will receive instruction (verbal and written) on recommended changes to diet and urinary habits to treat bladder pain for six (6) weeks before starting pelvic floor physical therapy.
  Interventions: Behavioral: Behavioral management; Other: Physical therapy

INTERVENTIONS:
Other: Acupuncture — traditional and electroacupuncture
  Arms: Acupuncture
Behavioral: Behavioral management — based on American urologic association guidelines
Other: Physical therapy — pelvic floor with biofeedback

SUMMARY:
The goal of this clinical trial is to learn if acupuncture in addition to behavioral changes can better treat in women with bladder pain syndrome (also known as interstitial cystitis) that have not received other treatments. The main question it aims to answer is:

Does acupuncture improve pain symptoms on the Interstitial Cystitis Index? Researchers will compare six (6) weeks behavioral management alone to behavioral management and acupuncture.

Participants will

* complete surveys about their bladder pain symptoms
* make behavioral changes that have been shown to improve bladder pain symptoms
* attend six (6) weekly acupuncture sessions
* attend six (6) weekly physical therapy sessions after finishing acupuncture

ELIGIBILITY:
Inclusion Criteria:

* Meets American Urologic Association (AUA) criteria for interstitial cystitis/bladder pain syndrome (IC/BPS): "An unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than 6 weeks duration, in the absence of other identifiable cause"
* Negative urine culture
* Has completed cystoscopic evaluation for IC/BPS

Exclusion Criteria:

* History of recurrent urinary tract infection (2 or more culture-positive in 6 months or 3 or more in 12 months)
* History of overactive bladder
* History of bleeding disorder or are currently on chronic anti-coagulation
* Post-void residual >100mL
* Has previously undergone any of the following treatments for any indication: acupuncture, pelvic floor physical therapy, pre-tibial nerve stimulation (PTNS), sacral neuromodulation, or intradetrusor Botox
* Prior bladder augmentation
* Currently undergoing or will undergo treatment for a urologic or gynecologic malignancy
* Currently pregnant (if applicable, based on self-report)
* Implanted pacemaker or defibrillator (AICD) or any metallic implants below umbilicus (eg hip or knee replacements)
* Non-English speaking and reading

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
O'Leary-Sant Interstitial Cystitis Index (OLSICI) | Baseline, every 2 weeks x3 (6 week study protocol period), every 4 weeks x 13 (52 week post-treatment period)
  Validated 8-item questionnaire with reported scores ranging 0-37. Higher scores are consistent with worse symptoms.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | x1 (end of 6 week study protocol period), x1 (end of 1 year post-treatment period)
  Validated 1-item likert-scale question on a scale from 1 (very much better) to 7 (very much worse).
Short Form (SF-36) | x1 (end of 6 week study protocol period), x1 (end of 1 year post-treatment period)
  Validated 36-item questionnaire. Higher scores are consistent with worse symptom control.
Genitourinary Pain Index (GUPI) | Baseline, every 2 weeks x3 (6 week study protocol period), every 4 weeks x 13 (52 week post-treatment period)
  Validated 9-item questionnaire with reported scores ranging 0-45. Higher scores are consistent with worse symptom control.
Number of additional treatments used during study period | 1 year post-treatment period
  Treatments include pharmacotherapy, intradetrusor botox, neuromodulation, cyclosporine
Number of unscheduled interactions | 1 year post-treatment period
  Unscheduled interactions include any phone calls, messages, or unplanned visits

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No